CLINICAL TRIAL: NCT05761548
Title: Study on the Development of Neonatal Cerebral Blood Flow Based on Ultrafast Ultrasound Doppler Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Liu Yunfeng, associate chief physician, Peking University Third Hospital
Other Study IDs: M2022211
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mature
  Interventions: Diagnostic Test: ultrafast ultrasound power Doppler imaging
- preterm
  Interventions: Diagnostic Test: ultrafast ultrasound power Doppler imaging

INTERVENTIONS:
Diagnostic Test: ultrafast ultrasound power Doppler imaging — ultrafast ultrasound power Doppler imaging for neonatal brain microvessels

SUMMARY:
Recently, with the development of perinatal medicine in China, the establishment of neonatal intensive care unit (NICU) and the improvement of respiratory support technology, the survival rate of preterm and term neonates has been significantly improved. However, the brain development of preterm neonates is incomplete compared with that of full-term neonates. Therefore, during the extrauterine cultivation of preterm neonates, clinical intervention should be carried out according to their brain development to achieve the same development status as that of full-term neonates. There are many clinical inspection methods to monitor the brain development of preterm neonates, such as EEG, functional near-infrared spectroscopy imaging, etc. However, these technologies cannot assess the brain development of premature infants systematically and completely. Because of the existence of neurovascular coupling, brain function and cerebral blood flow are closely related, so the detection of cerebral blood flow can reflect brain development and brain function. Ultrafast ultrasound power Doppler imaging technology is an emerging, real-time, high-resolution microvascular imaging technology. In this study, we first used ultrafast ultrasound power Doppler imaging technology to image the cerebral blood flow of preterm neonates at different gestational ages to evaluate the development of cerebral blood flow of preterm and term neonates and provide guidance for the clinical intervention of preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* neonates without cerebral diseases

Exclusion Criteria:

* neonates with cerebral diseases

Ages: 24 Weeks to 40 Weeks | Sex: All
Age Groups: Child
Study Population: From May 2022 to May 2023, newborns hospitalized in neonatal and NICU wards in the Peking University Third Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Intrauterine cerebral blood flow development of neonates | 30 min
Extrauterine cerebral blood flow development of neonates | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China